CLINICAL TRIAL: NCT04709198
Title: The Association Between Nutritional Status and Muscle Wasting and Fraility in Intensive Care Patients
Brief Title: Nutritional Status, Muscle Wasting and Fraility in Intensive Care Patients
Status: Completed | Type: Observational
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, Melda Kangalgil, Research Assistant, Karadeniz Technical University
Other Study IDs: 202057
Record Dates: First submitted 2021-01-04; First posted 2021-01-14 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Critical Illness; Nutritional Disorder
MeSH Terms: conditions — Critical Illness; Nutrition Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The risk of muscle wasting is high in the intensive care unit patients during the treatment process and this condition is associated with adverse clinical outcomes. The etiology of muscle wasting is multifactorial and medical nutrition therapy plays a key role in muscle wasting treatment and prevention. The aim of this study is assesing the malnutrition and fraility, anthropometric measurements, and muscle mass by ultrasound at the first admission to the intensive care unit and to determine the nutritional factors affecting clinical outcomes. In addition, it is planned to determine the risk factors affecting the change of anthropometric measurements and muscle wasting in the first week during the intensive care unit.

DETAILED DESCRIPTION:
A nutrition-focused physical examination is an integral component in the assessment of critically ill patients. Malnutrition, muscle wasting, and frailty are multidimensional clinical conditions in critically ill patients and are associated with adverse outcomes. Although malnutrition, muscle wasting and frailty are linked, the exact relation between them is unsure. As a result of evaluating these conditions together, it is planned to develop new treatment strategies and to improve the clinical results of patients by determining the relationship between medical nutrition therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥45 years and ≤80 years, male or female
* Expected ICU stay of seven days or longer
* Written informed consent or requirements of local/national ethical committee

Exclusion Criteria:

* Pregnancy or breastfeeding
* Neuromuscular conditions (e.g., multiple sclerosis, muscular dystrophy, spinal cord injury, Guillain-Barre syndrome)
* Terminal cancer
* Dialysis dependent chronic renal failure
* Intoxication
* Burn injury
* A cognitive impairment prior to the acute illness that is associated with admission to ICU that would impair capacity to follow verbal instructions
* Concurrent enrolment in a nutrition-related interventional study at the time of screening

Ages: 45 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Critically ill patients aged between 45-80 years of both sexes
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2020-10-20 (Actual); Primary Completion 2021-06-20 (Actual); Study Completion 2022-06-20 (Actual)

PRIMARY OUTCOMES:
Changes in muscle cross-sectional area | Baseline and 7 days
  Rectus femoris muscle cross-sectional area will be evaluated by ultrasound.
Changes in anthropometric measurements | Baseline and 7 days
  Triceps skinfold thickness will be measured by caliper.

SECONDARY OUTCOMES:
Duration of mechanical ventilation | Time of admission to the ICU until the time of discharge from the intensive care unit, up to 1 year
  Duration of mechanical ventilation in survivors and non survivors
Mortality rate | Time of admission to the ICU until the time of discharge from the intensive care unit, up to 1 year
  ICU mortality

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet Oguzhan Kucuk, MD, Principal Investigator — Karadeniz Technical University; Hulya Ulusoy, Professor, Principal Investigator — Karadeniz Technical University; Ayse Ozfer Ozcelik, Professor, Principal Investigator — Ankara University
Locations (1):
- Karadeniz Technical University Faculty of Health Sciences, Trabzon, Eyalet/Yerleşke, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No